CLINICAL TRIAL: NCT04654923
Title: Epidemiological Survey on Perioperative Hypersensitivity Reactions in France by the GERAP Network (Groupe d'étude Des réactions Anaphylactiques périopératoires)
Brief Title: GERAP's Epidemiological Survey on Perioperative Hypersensitivity Reactions
Acronym: SERAP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8038
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hypersensitivity, Drug
Keywords: anaphylaxis; perioperative; hypersensitivity reactions; neuromuscular blocking agents; hypnotics
MeSH Terms: conditions — Drug Hypersensitivity; Anaphylaxis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative hypersensitivity reactions are still associated with significant morbidity and mortality despite early recognition and use of epinephrine. The epidemiology of these reactions evolves over time and changes with clinical practice. The main objective is to study the epidemiology of these reactions over a 10-year period, including patient phenotype, reaction phenotype and outcome of the allergic work-up.

ELIGIBILITY:
Inclusion Criteria:

* Minor and major subject
* Subject having experienced a perioperative hypersensitivity reaction between January the 1st 2017 and December the 31st 2027.
* Referred for an allegro-anesthetic workup
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Inability to provide the subject with research information
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject having experienced a perioperative hypersensitivity reaction
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2031-05-12 (Estimated); Study Completion 2031-05-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of incidence of all perioperative hypersensitivity reactions referred in an allegro-anesthetic | Outcome is analysed every 2 years over a 10 years period

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Michel MERTES, MD, PhD, Study Director — Strasbourg University Hospitals - Anesthesia-intensive care unit; Charles TACQUARD, MD, Principal Investigator — Strasbourg University Hospitals - Anesthesia-intensive care unit
Locations (1):
- Service d'anesthésie-réanimation - CHU de Strasbourg - France, Strasbourg, France

REFERENCES:
- [Derived] Tacquard C, Serrier J, Viville S, Chiriac AM, Franchina S, Gouel-Cheron A, Giraudon A, Le Guen M, Le Quang D, Malinovsky JM, Petitpain N, Demoly P, Mertes PM; GERAP study group. Epidemiology of perioperative anaphylaxis in France in 2017-2018: the 11th GERAP survey. Br J Anaesth. 2024 Jun;132(6):1230-1237. doi: 10.1016/j.bja.2024.01.044. Epub 2024 Mar 16. PMID 38493055